CLINICAL TRIAL: NCT06190067
Title: Azacitidine Plus PD-1 Therapy for Relapsed/Refractory Hodgkin Lymphoma
Brief Title: Azacitidine Plus PD-1 Therapy for R/R Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liren Qian, Vice Director, Navy General Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA2023
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Relapsed Classic Hodgkin Lymphoma; Refractory Classic Hodgkin Lymphoma
MeSH Terms: interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacitidine Plus PD-1 therapy (Experimental): Patients were treated by Azacitidine plus PD-1 therapy
  Interventions: Drug: Azacitidine Plus PD-1 therapy

INTERVENTIONS:
Drug: Azacitidine Plus PD-1 therapy — Patients were treated by Azacytidine(75 mg/m2 subcutaneous injection qd on days 1-7) plus PD-1 therapy(200mg iv qd d8)
  Other Names: Azacitidine Plus PD-1 antibody

SUMMARY:
The goal of this phase 2 trial is to test the safety and efficacy of azacitidine when given together with PD-1 therapy in treating patients with relapsed/refractory classic Hodgkin lymphoma.

DETAILED DESCRIPTION:
The investigators will evaluate response rate, progression free survival (PFS), overall survival (OS), and toxicity of azacytidine combined with PD-1 therapy in classic relapsed/refractory Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Hodgkin Lymphoma according World Health Organization (WHO) classification.
* Patient is ≥ 18 years of age at the time of signing the informed consent form (ICF).
* Patient must understand and voluntarily sign an ICF prior to any study-specific assessments/procedures being conducted.
* Patient is willing and able to adhere to the study visit schedule and other protocol requirements.
* Relapsed (after partial or complete response) or refractory AITL after at least one line of systemic therapy (there is no mandatory resting period after the previous treatment as long as the biochemistry and hematology labs meet the inclusion criteria as below).
* Meet the following lab criteria: Absolute Neutrophil Count (ANC) ≥ 1,5 x 10^9/L (≥ 1 x 10^9/L if bone marrow (BM) involvement by lymphoma); Platelet ≥ 75 x 10^9/L (≥ 50 x 10^9/L if BM involvement by lymphoma); Hemoglobin ≥ 8 g/dL.
* Anticipated life expectancy at least 3 months.

Exclusion Criteria:

* Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment.
* Any instability of systemic disease, including but not limited to severe cardiac, liver, kidney, or metabolic disease need therapy.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  ORR was defined as the proportion of patients who achieved CR or PR as their best response

SECONDARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 2 year
  OS was defined as time from diagnosis to death from any cause or the last follow-up
Progression Free Survival (PFS) | 18 months
  PFS using local assessment of progressive disease according to Lugano Response Criteria (2014)

CONTACTS AND LOCATIONS:
Overall Officials: Liren Qian, PhD, Principal Investigator — Navy General Hospital, Beijing
Locations (1):
- Navy General Hospital, Beijing, Beijing Municipality, China